CLINICAL TRIAL: NCT06223048
Title: A Phase 2, Randomized, Open Label Study of AMDX-2011P as a Retinal Tracer in Participants With Primary Open Angle Glaucoma
Brief Title: A Study of AMDX-2011P in Participants With Primary Open Angle Glaucoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amydis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AMDX-2011P-202
Record Dates: First submitted 2023-12-14; First posted 2024-01-25 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Primary Open Angle Glaucoma
Keywords: POAG
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: Phase 2, randomized, parallel arm, open-label, masked endpoint study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMDX-2011P 50 mg (Experimental): AMDX2011P mg 50 (2ml) single bolus injection intravenous for diagnostic review
  Interventions: Drug: AMDX-2011P
- AMDX-2011P 100 mg (Experimental): AMDX2011P 100mg (4ml) single bolus injection intravenous for diagnostic review
  Interventions: Drug: AMDX-2011P

INTERVENTIONS:
Drug: AMDX-2011P — AMDX-2011P single bolus injection intravenous for diagnostic review

SUMMARY:
The purpose of this research study is to assess the ability of AMDX- 2011P to identify amyloid deposits in the retina of participants with Primary Open Angle Glaucoma (POAG).

DETAILED DESCRIPTION:
This open-label, masked endpoint assessment study will evaluate safety, tolerability, plasma pharmacokinetics (PK) and biological activity of intravenous (IV) doses of AMDX-2011P in participants with POAG. Assessments of retinal images will be conducted by centrally masked assessors.

Participants will be admitted to the study site where eye examination and retinal imaging will be conducted before administration of the study drug. AMDX-2011P will be administered through a single IV bolus injection followed by safety assessments, retinal imaging, and blood collection and PK.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of primary open angle glaucoma in both eyes
2. Able to fixate
3. Glaucomatous optic nerve damage in both eyes, as determined by an investigator as part of an eye exam

Exclusion Criteria:

1. Participants unable to read or write
2. Ocular media is not sufficiently clear to obtain acceptable quality images
3. Participants with presence of any ocular pathology other than glaucoma in the study eye (cataracts are acceptable)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
AMDX-2011P Adverse Events Profile | 8 days
  Incidence, nature and severity of AEs/SAEs

SECONDARY OUTCOMES:
Concentration of AMDX-2011P | 2 hours
  Plasma PK Concentration (CMax)
Pharmacokinetic Analysis of AMDX-2011P | 2 hours
  Area under the plasma versus time curve (AUC)
Biological Activity | 1 day
  Detection of amyloid deposits in the retina after intravenous AMDX-2011P administration using a conventional retinal fundus fluorescence imaging device.

CONTACTS AND LOCATIONS:
Overall Officials: David Bingaman, Study Director — Amydis Inc.
Locations (3):
- United States (3):
  - Associated Retina Consultants, Phoenix, Arizona
  - Global Research Management, Glendale, California
  - Eye Research Foundation, Newport Beach, California

IPD SHARING:
Plan to Share IPD: No